CLINICAL TRIAL: NCT06644599
Title: Integrated Proactive Wireless Monitoring for Clinical Deterioration: A Stepped Wedge Randomized Trial
Brief Title: Wireless Monitoring for Clinical Deterioration
Acronym: i-PROTECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Dr Yaseen Arabi, Chairman intensive care unit, King Saud Bin Abdulaziz University for Health Sciences
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ICT23R/006/08
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-09

CONDITIONS: Inpatient Facililty Diagnoses
Keywords: inpatients; wireless monitoring; mortality; cardiopulmonary failure

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be maintained with a research coordinator who is not involved in this trial, and the ward allocation will remain concealed from the research and clinical teams throughout the study and will be revealed for a given sequence only 1 month before the implementation of the intervention to allow training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Wireless monitoring (Active Comparator): Wireless monitoring will be applied on patients who are at high risk, identified as having a National Early Warning Score (NEWS)-2 score of 5 or higher, patients with lower NEWS-2 scores if the clinical team has a clinical concern, patients with Critical Care Response Team (CCRT) activation regardless of NEWS-2 score and post-ICU discharges regardless of NEWS-2 score. The technology allows to have alarms for patients who meet preset thresholds for vital signs. These alarms are transmitted through a mobile device to the charge nurse of the related ward. The wireless system will be monitored 24/7 by a critical care nurse
- Control (No Intervention): Usual care with no wireless monitoring.

INTERVENTIONS:
Device: wireless monitoring — The monitoring wireless system will continuously monitor the heart rate, oxygen saturation (SpO2), respiratory rate, and blood pressure and in selected patients electrocardiography (ECG).

SUMMARY:
The study evaluates whether implementing a wireless monitoring system for patients admitted to hospital wards reduces mortality and cardiopulmonary failure.

DETAILED DESCRIPTION:
The trial is designed as a stepped-wedge cluster RCT. Hospital wards (which constitute clusters in this design) will be randomized to have wireless monitoring, 7 wards at a time, with each 7 wards constituting a sequence. The study consists of 5 periods of two-month sequences followed by a one-month transition time with a phased introduction of the intervention. In the first period, all wards will have no wireless monitoring. After a baseline period of 2 (+1 washout) months, the intervention (monitoring system) will be implemented in a randomly selected new sequence every 3-month period until the intervention is implemented in all sequences.

ELIGIBILITY:
Inclusion Criteria:

Ward level Inpatient wards, defined as wards used to manage adult inpatients.

Patient level

1. Aged 14 years or older
2. Checked in as inpatient status to one of the study wards

Exclusion Criteria:

Ward level

1. Cardiology, pediatric, obstetric wards
2. ICUs and emergency departments
3. Operating rooms
4. Outpatient clinics
5. Daycare wards, endoscopy, outpatient procedure areas, hemodialysis units

Patient level No commitment for full life support at the time of arrival to the study ward (designated as Do-Not-Resuscitate status)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13160 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of 30-day in-hospital mortality, cardiac arrest, requirement of vasopressor or intubation | 30 days
  After hospital admission within 30 days

SECONDARY OUTCOMES:
Cardiac arrest | 30 days
  cardiac arrest within 30 days of hospital admission
Requirement of vasopressors | within 30 days of hospital admission
  use of vasopressors/inotropic support
Requirement of intubation | 30 days
  need for mechanical ventilation within 30 days of hospital admission
Hospital length of stay | 90 days
  censored at 90 days
Transfer to ICU | 30 days
  ICU admission within 30 days of hospital admission
ICU- free days | 30 days
  in the first 30 days of hospital admission
CCRT activation | 30 days
  Critical care response team activation within 30 days of hospital admission

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at the discretion of the Principal investigator

REFERENCES:
- [Background] Jones D, Mitchell I, Hillman K, Story D. Defining clinical deterioration. Resuscitation. 2013 Aug;84(8):1029-34. doi: 10.1016/j.resuscitation.2013.01.013. Epub 2013 Jan 31. PMID 23376502
- [Background] Buist M, Bernard S, Nguyen TV, Moore G, Anderson J. Association between clinically abnormal observations and subsequent in-hospital mortality: a prospective study. Resuscitation. 2004 Aug;62(2):137-41. doi: 10.1016/j.resuscitation.2004.03.005. PMID 15294398
- [Background] Al-Qahtani S, Al-Dorzi HM, Tamim HM, Hussain S, Fong L, Taher S, Al-Knawy BA, Arabi Y. Impact of an intensivist-led multidisciplinary extended rapid response team on hospital-wide cardiopulmonary arrests and mortality. Crit Care Med. 2013 Feb;41(2):506-17. doi: 10.1097/CCM.0b013e318271440b. PMID 23263618
- [Background] Arabi YM, Al-Dorzi HM, Alamry A, Hijazi R, Alsolamy S, Al Salamah M, Tamim HM, Al-Qahtani S, Al-Dawood A, Marini AM, Al Ehnidi FH, Mundekkadan S, Matroud A, Mohamed MS, Taher S. The impact of a multifaceted intervention including sepsis electronic alert system and sepsis response team on the outcomes of patients with sepsis and septic shock. Ann Intensive Care. 2017 Dec;7(1):57. doi: 10.1186/s13613-017-0280-7. Epub 2017 May 30. PMID 28560683
- [Background] Hogan H, Healey F, Neale G, Thomson R, Vincent C, Black N. Preventable deaths due to problems in care in English acute hospitals: a retrospective case record review study. BMJ Qual Saf. 2012 Sep;21(9):737-45. doi: 10.1136/bmjqs-2011-001159. PMID 22927487
- [Background] Armitage M, Eddleston J, Stokes T; Guideline Development Group at the NICE. Recognising and responding to acute illness in adults in hospital: summary of NICE guidance. BMJ. 2007 Aug 4;335(7613):258-9. doi: 10.1136/bmj.39272.679688.47. No abstract available. PMID 17673769
- [Background] Smith GB. In-hospital cardiac arrest: is it time for an in-hospital 'chain of prevention'? Resuscitation. 2010 Sep;81(9):1209-11. doi: 10.1016/j.resuscitation.2010.04.017. Epub 2010 Jul 2. PMID 20598425
- [Background] Weenk M, van Goor H, Frietman B, Engelen LJ, van Laarhoven CJ, Smit J, Bredie SJ, van de Belt TH. Continuous Monitoring of Vital Signs Using Wearable Devices on the General Ward: Pilot Study. JMIR Mhealth Uhealth. 2017 Jul 5;5(7):e91. doi: 10.2196/mhealth.7208. PMID 28679490
- [Background] Breteler MJM MSc, Huizinga E, van Loon K, Leenen LPH, Dohmen DAJ, Kalkman CJ, Blokhuis TJ. Reliability of wireless monitoring using a wearable patch sensor in high-risk surgical patients at a step-down unit in the Netherlands: a clinical validation study. BMJ Open. 2018 Feb 27;8(2):e020162. doi: 10.1136/bmjopen-2017-020162. PMID 29487076
- [Background] Breteler MJM, KleinJan EJ, Dohmen DAJ, Leenen LPH, van Hillegersberg R, Ruurda JP, van Loon K, Blokhuis TJ, Kalkman CJ. Vital Signs Monitoring with Wearable Sensors in High-risk Surgical Patients: A Clinical Validation Study. Anesthesiology. 2020 Mar;132(3):424-439. doi: 10.1097/ALN.0000000000003029. PMID 31743149
- [Background] Bellomo R, Ackerman M, Bailey M, Beale R, Clancy G, Danesh V, Hvarfner A, Jimenez E, Konrad D, Lecardo M, Pattee KS, Ritchie J, Sherman K, Tangkau P; Vital Signs to Identify, Target, and Assess Level of Care Study (VITAL Care Study) Investigators. A controlled trial of electronic automated advisory vital signs monitoring in general hospital wards. Crit Care Med. 2012 Aug;40(8):2349-61. doi: 10.1097/CCM.0b013e318255d9a0. PMID 22809908
- [Background] Subbe CP, Duller B, Bellomo R. Effect of an automated notification system for deteriorating ward patients on clinical outcomes. Crit Care. 2017 Mar 14;21(1):52. doi: 10.1186/s13054-017-1635-z. PMID 28288655
- [Background] Taenzer AH, Pyke JB, McGrath SP, Blike GT. Impact of pulse oximetry surveillance on rescue events and intensive care unit transfers: a before-and-after concurrence study. Anesthesiology. 2010 Feb;112(2):282-7. doi: 10.1097/ALN.0b013e3181ca7a9b. PMID 20098128
- [Background] Mdege ND, Man MS, Taylor Nee Brown CA, Torgerson DJ. Systematic review of stepped wedge cluster randomized trials shows that design is particularly used to evaluate interventions during routine implementation. J Clin Epidemiol. 2011 Sep;64(9):936-48. doi: 10.1016/j.jclinepi.2010.12.003. Epub 2011 Mar 16. PMID 21411284
- [Background] Porsdam Mann S, Savulescu J, Sahakian BJ. Facilitating the ethical use of health data for the benefit of society: electronic health records, consent and the duty of easy rescue. Philos Trans A Math Phys Eng Sci. 2016 Dec 28;374(2083):20160130. doi: 10.1098/rsta.2016.0130. PMID 28336803
- [Background] Gonzales R, Anderer T, McCulloch CE, Maselli JH, Bloom FJ Jr, Graf TR, Stahl M, Yefko M, Molecavage J, Metlay JP. A cluster randomized trial of decision support strategies for reducing antibiotic use in acute bronchitis. JAMA Intern Med. 2013 Feb 25;173(4):267-73. doi: 10.1001/jamainternmed.2013.1589. PMID 23319069
- [Background] van Wyk JT, van Wijk MA, Sturkenboom MC, Mosseveld M, Moorman PW, van der Lei J. Electronic alerts versus on-demand decision support to improve dyslipidemia treatment: a cluster randomized controlled trial. Circulation. 2008 Jan 22;117(3):371-8. doi: 10.1161/CIRCULATIONAHA.107.697201. Epub 2008 Jan 2. PMID 18172036